CLINICAL TRIAL: NCT07168460
Title: Social Working Dogs Support To Children With Problematic School Absence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Swedish University of Agricultural Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-01706-01; N2021-0022 (Other Grant/Funding Number: Agria/SKK research fund)
Record Dates: First submitted 2025-09-01; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Learning Development; Quality of Life; School Attendance
Keywords: problematic school absence; school attendance; learning achievement; quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social working dogs team (Experimental): Children are randomized to this social working dogs team to receive dog-assisted educational tasks such as reading.
  Interventions: Behavioral: Dog-assisted support
- Special education teachers team (Active Comparator): Children are randomized to this active control group to perform educational tasks with the support of special educational teachers.
  Interventions: Behavioral: Special education teacher support

INTERVENTIONS:
Behavioral: Dog-assisted support — Children in the intervention group received dog-assisted support for 30 minutes per session, twice per week for 10-12 weeks. The process began with children meeting school dog with dog handlers either at their home or at school. During the intervention, children had physical contact with dogs as much as they wished and on consideration of dogs' welfare. The dog handler carried out some pedagogical tasks, such as children reading to the dog while the dog was next to the child or when its head was on the child's lap. The dog handler documented the process of each session in a protocol filled in after each session and observed the children on their educational tasks.
  Arms: Social working dogs team
Behavioral: Special education teacher support — Children in the control group met special education teachers and received pedagogical tasks involving Swedish, mathematics, etc. Similar to the dog team, special education teachers documented the process and observed the performance of children's educational tasks.
  Arms: Special education teachers team

SUMMARY:
The purpose of this project is to investigate whether trained social service dogs can increase students' school attendance and school motivation, and ultimately contribute to students reaching the basic learning goals. Main research questions are:

1. What are the effectiveness and cost-effectiveness of having social service dogs support at schools to improve learning outcome and school attendance in students with problematic school absence?
2. What are the risks to the health and well-being of those social working dogs when they work in the school environment as well as the challenges in bringing dogs to the schools?

Researchers compared the intervention group which consisted of students supported by social working dogs, to the control group of students supported by special education teachers. Participants were assigned to each group randomly. Students from each group met the support teams for 30 minutes per session, twice per week for 10-12 weeks. During the intervention, children had physical contact with dogs as much as they wished and on consideration of dogs' welfare. The dog handler carried out some pedagogical tasks, such as children reading to the dog while the dog was next to the child or when its head was on the child's lap. The dog handlers documented the process of each session and observed the children on their educational tasks. Children in the control group met special education teachers and received pedagogical tasks involving Swedish, mathematics, etc. Similar to the dog team, special education teachers documented the process and observed the performance of children's educational tasks.

DETAILED DESCRIPTION:
The aim of this project is to investigate whether an intervention delivered by trained social working dog teams can increase school attendance among school-age children in grades 3-9, contribute to children achieving the basic learning goals, and improve health-related quality of life. The study design is an individually-randomized controlled trial with two arms - intervention and control. Randomization is conducted at the individual level within each school through lottery. Schools in Sweden were contacted by sending out flyers. Principals who wanted their schools to participate in the project contacted the project manager. The selection criteria for inclusion in the project are children from grades 3-9 with at least 15% absence from school during at least one semester, receiving no additional support.The criteria for exclusion are as follows: children who had 50%-100% absenteeism for more than a year; children who were severely allergic to dogs or who had previous negative experiences with dogs; and children from grades 1-3. Additionally, children who had previously participated in an intervention with a social working dog were excluded, as the potential impact on the results is unknown. Participation was voluntary, and written consent forms from both children and parents/ guardians were obtained. The study population includes school-age children from grades 3-9 in Sweden. A sample size of around 64 school-going children with a 1:1 allocation was allocated within the schools into control and intervention groups. Primary outcome data were collected at the following time points: T0 - pre-intervention (the whole semester before intervention), T1 - the whole semester during intervention, and T2 - the whole semester after intervention. Secondary outcome data were collected at T0 - pre-intervention, T1 - immediately post intervention, T2 - 3 months post intervention, and T3 - 6 months post intervention.

ELIGIBILITY:
Inclusion Criteria:

- Children from grades 3-9 with at least 15% absence from school during at least one semester and receiving no additional support.

Exclusion Criteria:

* Children who had 50%-100% absenteeism for more than a year
* Children who were severely allergic to dogs or who had previous negative experiences with dogs
* Children from grades 1-3
* Children who had previously participated in an intervention with a social working dog.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
School absenteeism | T0-The whole semester before intervention (5 months pre-intervention), T1-The whole semester during intervention (5 months during intervention), and T2 - The whole semester after intervention (5 months after intervention).
  Children's weekly school attendance (%) were retrieved from school registration records on children's attendance.
Learning achievement | T0-The whole semester before intervention (5 months pre-intervention), T1-The whole semester during intervention (5 months during intervention), and T2 - The whole semester after intervention (5 months after intervention).
  Children's attainment of basic learning goals was measured through grades obtained on two subjects: Swedish and Mathematics. Children were graded as pass (Godkänd) or fail (Undergodkänd) in Swedish and Mathematics. Data were retrieved through school reports.

SECONDARY OUTCOMES:
Children's health-rated quality of life (HRQOL) | T0 - pre-intervention, T1 - immediately post intervention, T2 - 3 months post intervention, and T3 - 6 months post intervention
  Children's health-rated quality of life (HRQOL) of both control and intervention classes was measured using the Child Health Utility 9 Dimensions (CHU9D), a generic preference-based HRQOL measure for use in children and youth.

CONTACTS AND LOCATIONS:
Overall Officials: Lena Lidfors, Doctorate in Ethology, Principal Investigator — Swedish University of Agricultural Sciences
Locations (1):
- Uppsala University & Swedish University of Agricultural Sciences, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
IDP sharing plan has not been decided as they are sensitive data, and that we need approval from our university GDPR and legal department to do so.